CLINICAL TRIAL: NCT02937766
Title: A Phase III, Single-Center, Open-labeled, Randomized Controlled Study Assessing Injection Pain of Preservative-free Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL) When Administered Via Subcutaneous Auto-injector vs Intramuscular Injection Via Needle and Syringe in Healthy Post-menopausal Women
Brief Title: Study Assessing Injection Pain of Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL) When Administered Via Subcutaneous Auto-injector vs Intramuscular Injection Via Needle and Syringe in Healthy Post-menopausal Women
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Sponsor elected to discontinue the study prematurely due to business reasons
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMAG-HPC-HPM-301
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-03

CONDITIONS: Assessing Injection Pain of Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL) in Healthy Post-menopausal Women
MeSH Terms: interventions — 17 alpha-Hydroxyprogesterone Caproate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): Subcutaneous (SQ) injection using an autoinjector weekly over 4 weeks (4 injections)
  Interventions: Drug: Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL)
- Treatment B (Active Comparator): Intramuscular injection (IM) using syringe and needle weekly over 4 weeks (4 injections)
  Interventions: Drug: Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL)

INTERVENTIONS:
Drug: Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL)
  Other Names: Makena SQ
  Arms: Treatment A
Drug: Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL)
  Other Names: Makena
  Arms: Treatment B

SUMMARY:
To demonstrate that Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL) delivered subcutaneously via auto-injector is associated with less pain as compared to intramuscular injections of Makena®

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects aged 50 to 75 years of age, inclusive, at Screening Visit.
2. Follicle stimulating hormone (FSH) levels greater than 40 mIU/mL.
3. Naturally or surgically postmenopausal with or without an intact uterus.

Exclusion Criteria:

1. Have history of or positive test results for HIV or hepatitis B or C.
2. A significant history or current evidence of chronic infectious disease, organ dysfunction especially cardiovascular, renal, or hepatic disorders or other medical condition.
3. Receiving or have received chronic opioid therapy within 12 months.
4. Unwilling to stop taking/using:

   * pain medication.
   * topical analgesic or anti-inflammatory treatment. Topical analgesics must be washed out by at least 72 hours in the areas to be treated before randomization.
5. History of alcohol abuse (regularly drinks > 4 units of alcohol per day; 8 oz. beer, 3 oz. wine, 1 oz. spirits) or prescription/illicit drug abuse in the last 12 months.
6. Currently taking any estrogen/progesterone hormone replacement therapy (HRT).
7. History of allergy or sensitivity to hydroxyprogesterone caproate, castor oil or any of the constituents of the study medications or history of any drug hypersensitivity or intolerance.
8. Poorly controlled diabetes (Hgb A1C >8).
9. Current or history of thrombosis or thromboembolic disorders.
10. Known or suspected breast cancer, other hormone-sensitive cancer or tumor, or history of these conditions within the last 5 years.
11. Any current or recent (within previous 12 months) vaginal bleeding.
12. Uncontrolled hypertension.
13. A chronic pain condition (i.e. chronic back pain) that may confound the assessments of injection pain.

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10-07 (Actual); Primary Completion 2017-01-06 (Actual); Study Completion 2017-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Singla, MD, Principal Investigator — Lotus Clinical Research, LLC
Locations (1):
- Lotus Clinical Research, LLC, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment A: Subcutaneous (SQ) injection using an autoinjector weekly over 4 weeks (4 injections)
  Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL)
- Treatment B: Intramuscular injection (IM) using syringe and needle weekly over 4 weeks (4 injections)
  Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL)
Period: Overall Study
Arm/Group | Treatment A | Treatment B
Started | 30 | 30
Completed | 23 | 30
Not Completed | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A | Treatment B | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 27 | 50
  >=65 years | 7 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (6.39) | 56.5 (4.23) | 57.9 (5.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Average Pain Intensity
Description: Comparison of average pain intensity associated with the administration of Makena® via subcutaneous autoinjector versus intramuscular injection (averaged over 4 visits).
  Score on a scale: 0 (No Pain) up to 10 (Worst Pain Imaginable)
Time Frame: 4 weeks
Population: The Comparison of Average Pain Intensity outcome was not analyzed. Pain assessments for participants included Adverse Events of Injection Site Pain reporting. 3 participants in Treatment Group A and 2 participants in Treatment Group B reported Injection Site Pain.
Measure: Number; unit: Participants with Injection Site Pain
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 30
Participants with Injection Site Pain | 3 | 2

2. Secondary Outcome: Clinician Assessment of Ease of Injection Technique
Description: Investigate the clinician's assessment of the ease of injection technique associated with the administration of Makena® via subcutaneous auto-injector versus intramuscular injection as measured by a categorical scale.
  Scores were as follows: completely dissatisfied = -3; mostly dissatisfied = -2, somewhat dissatisfied = -1, neither satisfied nor unsatisfied = 0, somewhat satisfied = 1, mostly satisfied = 2, completely satisfied = 3
Time Frame: 4 weeks
Population: Analysis population is comprised of all subjects who were randomized and received study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 30
units on a scale | 2.8 (0.43) | 2.3 (1.32)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority; p = 0.093, t-test, 2 sided; The t-test tested the hypothesis of no treatment difference between treatment groups; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.1 to 0.9], Standard Error of Mean 0.25

3. Secondary Outcome: Clinician Assessment of Ease of Drug Preparation
Description: Investigate the clinician's assessment of the ease of drug preparation associated with the administration of Makena® via subcutaneous auto-injector versus intramuscular injection as measured by a categorical scale.
  Scores were as follows: completely dissatisfied = -3; mostly dissatisfied = -2, somewhat dissatisfied = -1, neither satisfied nor unsatisfied = 0, somewhat satisfied = 1, mostly satisfied = 2, completely satisfied = 3
Time Frame: 4 weeks
Population: Analysis population is comprised of all subjects who were randomized and received study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 30 | 30
units on a scale | 2.8 (0.43) | 2.5 (1.14)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority; p = 0.234, t-test, 2 sided — The t-test tested the hypothesis of no treatment difference between treatment groups; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.2 to 0.7], Standard Error of Mean 0.22

ADVERSE EVENTS:
Time Frame: Approximately 66 days
Arm/Group | Treatment A | Treatment B
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/30
Other Adverse Events (participants affected / at risk) | 17/30 | 13/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=30) | Treatment B (N=30)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=30) | Treatment B (N=30)
Injection site pain (General disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 2 (2) | 0 (0)
Injection site nodule (General disorders) | 2 (2) | 0 (0)
Injection site paraesthesia (General disorders) | 0 (0) | 1 (1)
Injection site pruritis (General disorders) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (4)
Dizziness (Nervous system disorders) | 1 (1) | 1 (2)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 2 (3) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The Sponsor elected to discontinue the study prematurely due to business reasons. The only parameters analyzed for efficacy were Ease of Drug Preparation and Ease of Injection Technique.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No